CLINICAL TRIAL: NCT04977999
Title: Comparative Effects of Eccentric-driven Exercise on Measures of Muscle Function When Combined With Aquatic Plyometric Exercise
Brief Title: Effects of Combining Eccentric and Aquatic Based Exercise on Muscle Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Student graduated, study is terminated.
Sponsor: Brennan Thompson (Other)
Responsible Party: Sponsor-Investigator, Brennan Thompson, Co-Principal Investigator, Utah State University
Organization: Utah State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11903
Record Dates: First submitted 2021-07-21; First posted 2021-07-27 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hydrotherapy
Keywords: plyometrics; vertical jump; depth jump; muscle strength; muscle power; eccentric training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized parallel two group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric training (Active Comparator): Eccentron (BTE Technologies, Inc.) training
  Interventions: Other: Exercise
- Aquatic training (Experimental): Hydroworks aquatic training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both arms/conditions use varying forms of exercise as the intervention.

SUMMARY:
The study will compare the effects of eccentric resistance training versus eccentric training combined with aquatic plyometric training on muscle function outcomes.

DETAILED DESCRIPTION:
This study will use a parallel, randomized group design. Two groups will be randomly formed with one group comprising an eccentric only resistance training condition (experimental control) and the other comprising an eccentric combined with aquatic-based plyometrics condition (experimental). All subjects, regardless of group, will train on a multiple-joint eccentric machine one time per week for 7 weeks. The combined group will also perform an aquatic-based exercise session one time (on a separate day from the eccentric training) per week. Muscle function will be assessed via a battery of tests including jumps, sprints, and isometric and eccentric maximal strength.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 30 years

Exclusion Criteria:

* Currently doing resistance exercise > 3 times per month or aerobic exercise at or more than 30 min, 5 days per week.
* Any lower limb injuries or surgery within a year of the study
* If any of the subject's are too tall for the Eccentron machine (>76 inches tall)
* If any of the subject's eccentric strength is measured to be greater than 725 pounds during the first test of eccentric strength.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Countermovement jump | 7 weeks
  Participants will perform three maximal counter movement vertical jumps on a force platform. Participants will be instructed to stand on the platform with their feet shoulder width apart with their hands on their hips. Participants will be instructed to quickly lower themselves to a comfortable depth then immediately jump as high as possible while landing with their legs relatively straight (Crane et al., 2020). A successful countermovement jump attempt will be counted if the participant lands on the platform with both feet and does not take a step before jumping (Palmer et al., 2014). A 1-minute rest period will be provided between each jump attempt. Participants will be asked to perform three practice jumps with their hands placed on hips. Following the completion of practice jumps, participants will perform 3 trials of countermovement jumping on land and 3 trials while immersed in water at waist-depth.
Depth jump | 7 weeks
  Participants will perform three maximal-effort depth jumps from a height of 0.4 meters onto a force plate. Participants will be instructed to step straight off of the box without lowering themselves prior to falling, then to land and quickly jump as high as they can with minimal ground contact time. A successful jump attempt requires landing on the force plate with both feet both from the drop as well as from the rebound jump. A 1-minute rest period will be provided between each jump attempt.
Maximal isometric strength | 7 weeks
  Participants will be tested on a custom-made isometric mid-thigh pull (IMTP) device. This device consists of a force plate set onto an aluminum plate to which a bar is attached via chains, which are adjustable for height. The subject will be fitted with an over-the-shoulder vest which will be secured to straps fixed to the force plate. The straps will be adjusted so that the participant's knee angle is set within a range of 125-145°, and the hip angle in a range of 140-150°, as has been suggested to be optimal (Comfort et al., 2019). Participants will be instructed to stand on the plate with feet shoulder width apart, and then to move to a point where the slack is all out of the straps. To initiate the pull, participants will be instructed to drive their feet through the floor as hard and as fast as they can, while keeping their feet and upper body in position, starting on the signal, and not performing a countermovement prior to the pull.
Maximal eccentric strength | 7 weeks
  Eccentric muscle strength will be assessed via Eccentron (BTE Technologies, Inc., USA), a seated isokinetic dynamometer. . The pedals will move toward the participant in an alternating motion, so that each leg will work isolaterally in a repetitive manner. There will be a total of 12 maximal effort repetitions, six for each leg. For testing purposes, the speed of this motion will be set at 23 cycles per minute, which is defined as a moderate speed (Gordon et al., 2019).
40-m sprint | 7 weeks
  Participants will perform three maximal-effort 40-m sprints on a hard track surface in accordance with procedures outlined by (Gordon et al., 2019). Sprint time will be measured by timing gates (Dashr Motion Performance Systems, Dashr LLC, Lincoln, Nebr., USA) positioned at the start and end points of the run distance. Participants will be instructed to start in a 3-point stance with their feet staggered and one hand on the ground. For the three point stance, participants will be instructed to place the front of their lead foot on a line 30 cm behind the start line, and to place the opposite hand of the lead foot on the starting line (Rimmer & Sleivert, 2000). The sprint will be started with the use of a verbal command and participants will be instructed to run through a line 10 meters past the second timing gate to ensure they give full effort throughout the entire measured distance. Three trials of sprints will be performed, with a rest period of two minutes between each trial.

SECONDARY OUTCOMES:
Muscle soreness | 7 weeks
  local muscle soreness will be assessed throughout the duration of the intervention period using a Wagner force algometer.
Muscle soreness (visual analog scale) | 7 weeks
  During the course of the training period, soreness levels will be assessed using a visual analog scale (VAS), in accordance with our previous procedures (Crane et al., 2020). The VAS will be administered at baseline (prior to the first training session) and for five consecutive days following the first training session of the first experimental week and then on three nonconsecutive, non-training days per week for the remaining six weeks (Crane et al., 2020).
Inertial measurement unit | 7 weeks
  3-axis microelectromechanical systems (MEMS) accelerometers (Blue Trident, Vicon Motion Systems) to assess center of mass during countermovement jumps

CONTACTS AND LOCATIONS:
Overall Officials: Brennan J Thompson, PhD, Study Chair — Utah State Univeristy
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No